CLINICAL TRIAL: NCT06758310
Title: Effects of an Individualized Exercise Program on Physical Performance Measures in Southwest Native American Adolescents
Brief Title: Exercise Effects in Native American Adolscents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Midwestern University (Other)
Responsible Party: Principal Investigator, Joshua Subialka, Assistant Professor, Midwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-24-0013
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Fitness Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Individualized exercise (Experimental)
  Interventions: Other: Individualized Exercise

INTERVENTIONS:
Other: Individualized Exercise — Each participant will be prescribed an individualized exercise program related to their fitness testing results and personal interests.

SUMMARY:
This longitudinal study will investigate effects of exercise participation in Southwest Native American adolescents, ages 11-17, from the Gila River Indian Community. Vital signs, physical activity participation adherence, physical performance measures, and psychological/social measures will be assessed. Participants will attend one educational presentation for the initial session, explaining the benefits of physical exercise and expectations throughout the program. Baseline measurements for strength, flexibility, and cardiovascular fitness will be taken as well as height, weight and blood pressure. Based on individual performance measures, each participant will be provided a personalized exercise program to complete 3-4 times/week for the duration for the duration of the study. Participants will also be provided an exercise journal to track their adherence to their exercise program each week. At the end of the session parents and adolescents separately will be asked to complete a written survey assessing physical, emotional, social, and school function. Physical performance measures will be taken every other week from the initial education and data collection session through 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Active members of the Gila River Indian Community (GRIC) with Native American ancestry
* Ages 11-17

Exclusion Criteria:

* Not active members of the GRIC or no Native American ancestry
* Age <11 or >17

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-11-16 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Push ups | 6 weeks
  Performed in 1 min
Sit ups | 6 weeks
  Performed in 1 min
Sit and Reach | 6 weeks
  Flexibility assessment
1 mile run | 6 weeks
  For time
Resting Heart Rate | 6 weeks

SECONDARY OUTCOMES:
Blood Pressure | 6 weeks

IPD SHARING:
Plan to Share IPD: No